CLINICAL TRIAL: NCT04779944
Title: Impact of SARS-CoV-2 Pandemic on Psychological State of Health Care Workers
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba A Yassa, Professor of Forensic Medicine and Clinical Toxicology, Assiut University
Other Study IDs: AssiutU1235
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: other — questionnaire
  Other Names: questionnaire

SUMMARY:
In COVID-19 pandemic, many health-care workers (HCWs) have worked in high-pressure environments. They have been exposed to and faced moral dilemmas in addition to infection exposure risk are increasing the risk of mental health disorders.

DETAILED DESCRIPTION:
Throughout the SARS-CoV-2 pandemic, many HCWs have worked in high-pressure environments. Moreover, they may have been exposed to trauma and/or faced moral dilemmas relating to challenges in the delivery of high-quality care, possibly due to a lack of experience or equipment, or as a result of low staffing levels. These unfavorable circumstances and exposure risk to infection are likely to increase the risk of mental health disorders such as post-traumatic stress disorder (PTSD) or depression, other anxiety disorders, substance misuse and suicide In the present study, This study aimed to assess the psychological state of HCWs who were facing challenges of SARS-CoV-2pandemic comparing them to non medical staff group based on use of the Hamilton Anxiety and Depression Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* All health workers team

Exclusion Criteria:

* no exclusion criteria

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All that work in the hospitals either doctors, nurses, dentist, pharmacysit
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire to assess the psychological impacts of SARS-CoV-2 on health care workers | 4 month
  Impact of SARS-CoV-2 on the Psychology of health care workers

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed Hussein, Principal Investigator — Assiut university- professor; Noha Abo Elfetoh, Study Chair — Assiut university- professor; Hoda Makhlouf, Study Chair — Assiut university- professor; Nahed Makhlouf, Study Chair — Assiut university- professor; Ahmed AbdelBaqy, Study Chair — Assiut university- Assistant professor; Heba Yassa, Study Director — Assiut university- professor
Locations (1):
- heba Yassa, Asyut, Egypt

REFERENCES:
- [Background] Williamson V, Stevelink SAM, Greenberg N. Occupational moral injury and mental health: systematic review and meta-analysis. Br J Psychiatry. 2018 Jun;212(6):339-346. doi: 10.1192/bjp.2018.55. PMID 29786495
- [Result] Li R, Pei S, Chen B, Song Y, Zhang T, Yang W, Shaman J. Substantial undocumented infection facilitates the rapid dissemination of novel coronavirus (SARS-CoV-2). Science. 2020 May 1;368(6490):489-493. doi: 10.1126/science.abb3221. Epub 2020 Mar 16. PMID 32179701
- [Result] Greenberg N, Docherty M, Gnanapragasam S, Wessely S. Managing mental health challenges faced by healthcare workers during covid-19 pandemic. BMJ. 2020 Mar 26;368:m1211. doi: 10.1136/bmj.m1211. No abstract available. PMID 32217624
- [Result] Brooks S, Amlot R, Rubin GJ, Greenberg N. Psychological resilience and post-traumatic growth in disaster-exposed organisations: overview of the literature. BMJ Mil Health. 2020 Feb;166(1):52-56. doi: 10.1136/jramc-2017-000876. Epub 2018 Feb 2. PMID 29420257